CLINICAL TRIAL: NCT00981448
Title: Nutrigenomics of Zinc Supplementation in Insulin Secretion and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Alan Shuldiner, Associate Dean for Personalized Medicine; Director, Program in Personalized and Genomic Medicine; Head, Division of Endocrinology, Diabetes and Nutrition, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00040355; 1KL2RR025006-01 (NIH)
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Diabetes
Keywords: zinc; diabetes; genetics
MeSH Terms: conditions — Diabetes Mellitus | interventions — Zinc Acetate; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zinc supplement (Experimental)
  Interventions: Dietary Supplement: Zinc acetate

INTERVENTIONS:
Dietary Supplement: Zinc acetate — 50mg of elemental zinc to be administered 2 times daily orally for 14 days.
  Other Names: Orazinc

SUMMARY:
The purpose of this study is to evaluate the effect of zinc supplementation on insulin secretion by genotype of SLC30A8.

DETAILED DESCRIPTION:
As diabetes increases at an alarming rate, strategies for prevention of this disease must be developed. For a given individual, there are both biologic (e.g., genetic) and environmental (e.g., lifestyle) factors that comprise her individual risk of diabetes. Researchers can take advantage the accumulating knowledge of these individual factors to design individualized strategies for diabetes risk assessment and prevention. For example, a mutation in a particular gene, SLC30A8, which encodes a zinc transporter, has been shown to increase the risk of diabetes probably through impairment of insulin secretion. In the proposed research project, the investigators aim to conduct a pilot study to see the effect of zinc supplementation on insulin secretion in people with and without this genetic mutation to see if zinc can improve insulin secretion in those with the mutation. The results from this study will help the investigators to plan a larger, more definitive study to determine if zinc supplementation can be used to prevent or treat diabetes in those with this mutation in SLC30A8.

ELIGIBILITY:
Inclusion Criteria:

* aged 21-70 years
* Amish decent
* genotyping of rs13266634 of SLC30A8 gene
* previously consented to contact for future studies and future use of DNA

Exclusion Criteria:

* Subject is a first-degree relative of another subject with the same SLC30A8 genotype
* diabetes mellitus (by history, treatment or random BG>200 mg;dl)
* gastrointestinal disease causing nausea, vomiting, or diarrhea including inflammatory bowel disease by history.
* rheumatoid arthritis by history
* albumin < 3.5 g/dL
* hemochromatosis by history
* hematocrit <34%
* liver disease by history
* alanine aminotransferase or aspartate aminotransferase greater than 2.5 times normal
* renal failure by history
* estimated glomerular filtration rate < 60 mL/min by MDRD equation
* use of thiazide diuretic and unwilling to discontinue if deemed safe in the opinion of the treating physician and study physician for 1 week prior to protocol initiation
* use of systemic corticosteroid and unwilling to discontinue if deemed safe in the opinion of the treating physician and study physician for 1 week prior to protocol initiation
* use of highly-active antiretroviral medications
* use of antipsychotic medications
* use of quinolone antibiotics
* use of tetracycline antibiotic and unwilling to discontinue if deemed safe in the opinion of the treating physician and study physician for 1 week prior to protocol initiation
* use of chelation therapy in the past month
* unwilling to withdraw from supplements for 1 week prior to the study and throughout study
* abnormal thyroid stimulating hormone (TSH) level
* serious disease precluding participation
* reported pregnancy or positive urine hCG test
* cancer diagnosis in past 2 years
* breastfeeding
* use of denture adhesive

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in acute insulin response from IVGTT. | 14 days

SECONDARY OUTCOMES:
change in insulin sensitivity | 14 days
change in disposition index | 14 days
self-report of history of symptoms of anemia or gastrointestinal symptoms during study | 14 days
change in serum zinc | 14 days
change in urinary zinc | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Shuldiner, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

REFERENCES:
- [Derived] Maruthur NM, Clark JM, Fu M, Linda Kao WH, Shuldiner AR. Effect of zinc supplementation on insulin secretion: interaction between zinc and SLC30A8 genotype in Old Order Amish. Diabetologia. 2015 Feb;58(2):295-303. doi: 10.1007/s00125-014-3419-1. Epub 2014 Oct 28. PMID 25348609